CLINICAL TRIAL: NCT02262416
Title: A Prospective Randomised Controlled Trial of GnRH Agonist and Progesterone Versus Progesterone Only for Luteal Phase Support in Antagonist Cycles
Brief Title: GnRH Agonist and Progesterone Versus Progesterone Only for Luteal Phase Support in Antagonist Cycles
Acronym: GALA
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Queensland Fertility Group (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 01102014
Record Dates: First submitted 2014-10-07; First posted 2014-10-13 (Estimated); Last update posted 2014-10-13 (Estimated); Status verified 2014-10

CONDITIONS: Infertility
Keywords: GnRH agonist; IVF
MeSH Terms: conditions — Infertility | interventions — Leuprolide

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- controls (Placebo Comparator): Normal saline of equivalent volume
- case (Active Comparator): 0.5mg Leuprolide acetate injection
  Interventions: Drug: leuprolide

INTERVENTIONS:
Drug: leuprolide — normal saline
  Other Names: lucrin
  Arms: case

SUMMARY:
In-Vitro Fertilisation (IVF) is the term commonly applied to a form of treatment for infertility that involves controlled ovarian hyperstimulation, egg maturation, egg collection, fertilisation, embryo culture and finally embryo transfer. The period after egg collection is called luteal phase. In Australia, vaginal progesterone is routinely used to support the lining of the uterus so that it is susceptible to implantation of the embryos.

More recently, there has been some suggestion that additional supplementation of luteal phase with GnRH agonist increases clinical pregnancy and live birth rate. These studies are however heterogeneous and results were inconsistent.

This study is a prospective randomised controlled trial of additional GnRH agonist in luteal phase of antagonist cycle. The primary hypothesis is that GnRH agonist increases the number of live birth . The secondary hypothesis is that this increases the clinical pregnancy rate, on-going pregnancy rate, without affecting the miscarriage rate, ovarian hyperstimulation rate and multiple pregnancy rate.

DETAILED DESCRIPTION:
In-vitro fertilization has been used since 1978 to treat women with infertility. It involves controlled ovarian stimulation, egg maturation, egg collection, fertilization and embryo culture and finally embryo culture. The luteal phase is the latter phase of the menstrual cycle which begins with the formation of the corpora lutea and ends in either pregnancy or luteolysis. The main hormone associated with this stage is progesterone, which is significantly higher during the luteal phase than other phases of the cycle. In the IVF setting, however, luteal phase deficiency is present and over the last 40 years various regimens have been used to support luteal phase of the cycle. Progesterone is currently widely used for this purpose and has shown to be effective in improving pregnancy and live birth rate (Van der Linden 2011).

There have been various other regimen used for luteal support in an attempt to further enhance luteal phase support such as oestrogen, HCG and GnRH agonist. The recent Cochrane study showed a significant benefit from addition of GnRH agonist to progesterone versus progesterone alone for the outcomes of live birth, clinical pregnancy and ongoing pregnancy. (Van Der Linden 2011) However, the conclusion derived from the metaanalysis were derived from limited number of studies that used various types additional luteal phase support, which also included a myriad of agonist and antagonist IVF cycles. Only ICSI cycles were included in the antagonist cycles.

A gonadotropin-releasing hormone (GnRH) agonist is a synthetic peptide that interacts with the GnRH hormone receptor to elicit its biologic response, the release of the pituitary hormones, FHS and LH. The exact mechanism of how GnRH could potentially increase pregnancy rate is unknown. Tesarik et al performed a randomised study in which addition of GnRH agonist increases implantation rate in donor recipient discounted the theory that GnRH acted on corpora lutea. It is suggested that GnRH acts directly on embryo to secrete BHCG hence enhances implantation. A prospective randomised study that was performed by Isik et al showed a promising result of use of GnRH agonist administration in the luteal phase of GnRH antagonist cycle (n=164). In this study, cases received 0.5mg leuprolide acetate in addition to 600mg micronised progesterone day 6 after ICSI compared to control group who received micronisd progesterone only. The study showed clinical pregnancy rate of 40% in cases vs 20% in control group. The increased number of multiple pregnancies in these studies could be partly explained by multiple embryos transferred. Answer is needed to determine if multiple pregnancy rate is higher if single embryo transfer is executed.

The studies performed by Tesarik et al and Isik et al showed promising increase in live birth rate and clinical pregnancy rates in antagonist cycles. Both studies were performed in clinical settings that were vastly different from Australia: multiple embryos were transferred, multiple luteal phase support were used in addition to progesterone and multiple pregnancy rates were high. Given the significant increase in pregnancy rate (>10%) were observed in these studies, if the increase is real, a RCT in Australia setting is needed prior to implementation of this intervention.

ELIGIBILITY:
Inclusion Criteria:

1. Single embryo transfer
2. Antagonist cycle with HCG trigger
3. Use of progesterone as luteal phase support (crinone or progesterone pessary )
4. Women undergoing their first IVF cycle with TFC
5. Age 18-42 inclusive

Exclusion Criteria:

No or frozen embryo transfer planned b. Use of other luteal support c. Known contraindication to the use of GnRH analogue

Ages: 18 Years to 42 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 200 (Estimated)
Dates: Start 2015-01; Primary Completion 2016-01 (Estimated); Study Completion 2016-01 (Estimated)

PRIMARY OUTCOMES:
live birth | 1 year
  live birth
on-going pregnancy | 3 months
  +ve fetal heart rate at nuchal scan

SECONDARY OUTCOMES:
pregnancy | 2 weeks
  positive serum pregnancy test
Ovarian hyperstimulation syndrome | 3 months
  hospitalisation due to the condition

CONTACTS AND LOCATIONS:
Locations (1):
- Queensland Fertility Group, Brisbane, Queensland, Australia

REFERENCES:
- [Background] Isik AZ, Caglar GS, Sozen E, Akarsu C, Tuncay G, Ozbicer T, Vicdan K. Reprod Biomed Online. 2009 Oct;19(4):472-7. Single-dose GnRH agonist administration in the luteal phase of GnRH antagonist cycles: a prospective randomized study. Medsafe New Zealand. www.medsafe.govt.nz/profs/datasheet/l/Lucrininj.pdf Tarlatzis BC, Bili H.Expert Opin Drug Saf. 2004 Jan;3(1):39-46. Safety of GnRH agonists and antagonists Tesarik J, Hazout A, Mendoza C.Hum Reprod. 2004 May;19(5):1176-80. Enhancement of embryo developmental potential by a single administration of GnRH agonist at the time of implantation Tesarik J, Hazout A, Mendoza-Tesarik R, Mendoza N, Mendoza C. Hum Reprod. 2006 Oct;21(10):2572-9. Beneficial effect of luteal-phase GnRH agonist administration on embryo implantation after ICSI in both GnRH agonist- and antagonist-treated ovarian stimulation cycles. Van der Linden M, Buckingham K, Farquhar C, Kremer JA, Metwally M.Cochrane Database Syst Rev. 2011 Oct 5;(10). Luteal phase support for assisted reproduction cycles